CLINICAL TRIAL: NCT01800019
Title: The Canadian HIV Quit Smoking Trial: Tackling the Co-morbidities of Depression and Cardiovascular Disease in HIV+ Smokers
Acronym: CANQUIT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2011824-01H; CTN 269 (Other Grant/Funding Number: CIHR Research Operating Grant)
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: HIV; Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy; Nicotine; Nicotine Chewing Gum; Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- NRT arm (Active Comparator): Drug: Nicotine Replacement Therapy (Nico-Derm® and Nicorette®)
  Dose: 7mg - 42mg depending on # of cigarettes smoked per day at study baseline, and withdrawal symptoms.
  Mode of Administration: Transdermal Patch
  Duration of Treatment: up to 24 Weeks
  Additionally, participants will be provided with a supply of short-acting nicotine gum in order to supplement their long acting NRT patch regimen.
  Individuals who smoke their first cigarette more than 30 minutes after waking are advised to use the 2 mg NRT gum. Participants who smoke their first cigarette within 30 minutes of waking will be advised to use the 4 mg NRT gum. Both NRT gum dosages will be recommended for use on an ad lib basis to address cravings and/or withdrawal symptoms, up to a maximum of 12 pieces of NRT gum per day.
  Interventions: Drug: Nicotine Replacement Therapy (NRT)
- NRT and HIV Tailored Quit Smoking Counseling (Active Comparator): Drug: Nicotine Replacement Therapy (Nico-Derm®)
  Dose: 7mg - 42mg depending on # of cigarettes smoked per day at study randomization and withdrawal symptoms.
  Mode of Administration: Transdermal Patch
  Duration of Treatment: up to 24 Weeks
  HIV tailored Smoking Cessation Counseling: The counseling consists of face-to-face sessions with a trained smoking cessation counselor at the start of the study, on your chosen quit date, and then at weeks 4, 8, 12 and 24; supportive telephone calls if needed.
  Interventions: Drug: Nicotine Replacement Therapy (NRT); Behavioral: HIV Tailored Quit Smoking Counseling
- Varenicline (VR) Arm (Active Comparator): Drug: Varenicline (Champix®)
  Doses: 0.5 mg once daily for 3 days(i.e.day 1-3 of the week prior to quit date) 0.5 mg twice daily for 4 days i.e. day 4-7) and 1 mg twice daily for the remainder of the treatment period
  Mode of Administration: Oral
  Duration of Treatment: 24 Weeks (+ 1 Week of Dose Escalation, total of 25 weeks)
  Interventions: Drug: Varenicline
- Varenicline (VR) and HIV Tailored Quit Smoking Counseling (Active Comparator): Drug: Varenicline (Champix®)
  0.5 mg once daily for 3 days(i.e.day 1-3 of the week prior to quit date) 0.5 mg twice daily for 4 days i.e. day 4-7) and 1 mg twice daily for the remainder of the treatment period
  Mode of Administration: Oral
  Duration of Treatment: 24 Weeks (+ 1 Week of Dose Escalation, total of 25 weeks)
  Intervention: HIV tailored Smoking Cessation Counseling: The counseling consists of face-to-face sessions with a trained smoking cessation counselor at the start of the study, on your chosen quit date, and then at weeks 4, 8, 12 and 24; supportive telephone calls if needed.
  Interventions: Drug: Varenicline; Behavioral: HIV Tailored Quit Smoking Counseling

INTERVENTIONS:
Drug: Nicotine Replacement Therapy (NRT)
  Other Names: Nico-Derm®; Nicoderm; the patch; Nicorette®; the gum
  Arms: NRT and HIV Tailored Quit Smoking Counseling; NRT arm
Drug: Varenicline
  Other Names: Champix
  Arms: Varenicline (VR) Arm; Varenicline (VR) and HIV Tailored Quit Smoking Counseling
Behavioral: HIV Tailored Quit Smoking Counseling — A cognitive behavioral therapy (CBT) oriented smoking cessation program tailored to HIV positive individuals.
  People Living with HIV/AIDS (PHA) tailored Canadian HIV Quit Smoking Counseling Intervention. It consists of face-to-face counseling sessions with a trained smoking cessation counsellor at randomization, on the identified quit date, and then at weeks 4, 8, 12, and 24.
  Other Names: Ottawa Model for Smoking Cessation
  Arms: NRT and HIV Tailored Quit Smoking Counseling; Varenicline (VR) and HIV Tailored Quit Smoking Counseling

SUMMARY:
The objectives of this trial are:

Primary objectives:

1. To determine among HIV+ individuals whether varenicline or NRT is more effective at helping individuals remain abstinent from smoking tobacco.
2. To determine among HIV+ individuals whether varenicline or NRT has the lowest side-effect profile.
3. To determine if the HIV tailored Quit Smoking Counselling Intervention, plus smoking cessation drug therapy, improves smoking cessation rates compared to smoking cessation drug therapy alone with usual care.

Secondary objective:

1. To determine whether the use of varenicline/NRT is safe in HIV+ patients who exhibit depressive symptoms.

Hypothesis:

That varenicline will result in higher quit smoking rates and that NRT will result in a lower side effect profile. Further, the HIV tailored quit smoking intervention will result in higher rates of smoking cessation over and above the pharmacological treatment alone. And finally, varenicline will be safe to use for HIV + individuals who exhibit depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. HIV positive
2. Adult (aged 18 or older)
3. Current smoker (more than 5 cigarettes per day)
4. Willing to set a date to quit smoking within the next 2-4 weeks
5. Currently on ART with an undetectable HIV viral load
6. Able to read/speak English or French
7. Able to provide written, informed consent as approved by the Ottawa Health Science Network Research Ethics Board and REBs at participating HIV clinic sites

Exclusion Criteria:

1. Contraindications to nicotine replacement therapy such as allergy to adhesive, serious cardiac arrhythmias (e.g., tachycardia), or vasospastic disease (e.g., Buerger's disease, Prinzmetal's variant angina)
2. Contraindications to varenicline such as hypersensitivity to varenicline or to any ingredient in the formulation or component of the container.
3. Reported previous severe intolerances to nausea or gastrointestinal symptoms.
4. Pregnant, lactating or planning to become pregnant during the study period or refuses a serum beta-HCG test.
5. Current severe renal impairment or currently taking Cimetidine
6. Previous or current seizure disorder and/or is taking anti-epileptic drugs
7. Psychosis and/or is taking anti-psychotic drugs
8. Diagnosed with severe major depressive episode requiring hospitalization within the past 12 months, previous psychiatric inpatient admission for any cause within the past 12 months, suicide attempt within the past 12 months active or current suicidal ideations as assessed by the BDI-II.
9. Current use of bupropion, varenicline or any nicotine replacement therapy.
10. Use of substances (e.g., crack cocaine) that would interfere with a participant's ability to adhere to the study schedule; determined by site coordinator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Smoking Status | at week 48
  The primary study end-point will be seven-day self-reported abstinence, and four week continuous abstinence rates at week 48, confirmed by expired carbon monoxide levels measured using a piCO+ Smokerlyzer (Smoke free defined as exhaled CO < 10 ppm). Study participants who are lost to follow-up (e.g., study drop-outs and those unavailable for follow-up) will be considered as smokers for the purposes of outcome analyses.

SECONDARY OUTCOMES:
Smoking Status: self report | quit date, weeks 4,8,12,16,20,24 and 48
  Seven-day point-prevalence, and 4-week continuous abstinence(if time interval permits), assessed by self-report and by expired carbon monoxide levels measured using a piCO+ Smokerlyzer.
  In addition, self-reported 4-week continuous abstinence rates (CAR) will be reported.
Smoking status: CO expired | randomization, quit date, 4, 8, 12, 16, 20, 24
  Smoke free status will be objectively measured by exhaled CO levels (<10ppm) with a Bedfont Smokerlyzer instrument.
Smoking cessation treatment integrity and patient satisfaction | Baseline through Week 48
  Study Medication: Adherence to NRT and varenicline will be assessed by participant self-reported adherence to medication at each study visit.
  Counseling Intervention: Each clinic site will have an HIV clinic health care provider who will be trained in administering the standardized HIV quit smoking intervention.
  Program Satisfaction Form will be completed by all study participants at the end of the study. At post-quit dates, treatment adherence will be assessed by a self-report measure of the amount of NRT or varenicline taken, number of cigarettes smoked in the previous 7 days, and marked changes in mood.
  Study coordinator will assess rates of discontinuation of varenicline or NRT. Participants who discontinue varenicline or NRT will still be followed according to the original schedule.
Behavioral-Psychosocial | Baseline to Week 48
  * The Minnesota Nicotine Withdrawal Scale
  * The Center for Epidemiological Studies Depression Scale
  * Smoking Self-Efficacy Questionnaire
  * EuroQol(EQ-5D)This scale is a brief, standardized, generic measure of HR-QOL that provides a 5-item profile of patient function and a global health state rating
  * Beck Depression Inventory
  * Experiences in Close Relationships
  * Stages of Change Questionnaire
  * Adherence to Treatment Questionnaire
  * Life Events Questionnaire
  * Use of Cessation Resources Survey
Cardiovascular Parameters | From baseline through 48 weeks
  The following parameters will be compared:
  1. Weight
  2. Height
  3. Waist circumference (defined by Heart and Stroke Foundation)
  4. Blood pressure
Immune Function | 12, 24, and 48 weeks
  Changes in:
  1. CD4-T-lymphocyte count and percentage
  2. HIV viral load
  3. CD8-T-lymphocyte count and percentage

CONTACTS AND LOCATIONS:
Overall Officials: Louise Balfour, PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273